CLINICAL TRIAL: NCT00962403
Title: Evaluation of a Yoga Intervention for Post-Traumatic Stress Disorder
Acronym: EYIPTSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Sat Bir Khalsa, PhD, Study Principal Investigator, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2009-P-000717; 08144033
Record Dates: First submitted 2009-08-13; First posted 2009-08-20 (Estimated); Last update posted 2013-03-20 (Estimated); Status verified 2013-03

CONDITIONS: Post-Traumatic Stress Disorder
Keywords: post traumatic stress disorder; yoga; meditation; military; veteran; trauma; stress; depression; anxiety; insomnia; autonomic
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Wounds and Injuries; Depression; Anxiety Disorders; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Yoga treatment (Experimental)
  Interventions: Behavioral: Yoga treatment
- Waitlist (No Intervention): Waitlist control, no active treatment, treatment as usual, active treatment offered after waitlist control period. This study began as a single arm treatment trial and then transitioned to a randomized controlled trial.

INTERVENTIONS:
Behavioral: Yoga treatment — The 10-week Kripalu-style yoga treatment will consist of 20 biweekly 90-minute group training/practice sessions. In addition, subjects will also receive CD's and written instructions for the daily 15-minute sessions, which they will use to guide them through the yoga procedures to be done at home.
  Other Names: Kripalu Yoga
  Arms: Yoga treatment

SUMMARY:
The main objective of this preliminary randomized controlled clinical trial is to establish efficacy and feasibility of a yoga-based treatment for PTSD in military veterans as compared to a delayed yoga treatment (waitlist control) group. Secondary objectives are to evaluate PTSD characteristics that may also be improved with the treatment and acceptability and compliance with the treatment.

DETAILED DESCRIPTION:
Specific Aims:

1. To evaluate the hypothesis that a 10-week yoga-based intervention will reduce PTSD severity to a statistically and clinically significant degree relative to a pretreatment baseline evaluation and to a waitlist control group.
2. To evaluate the hypothesis that PTSD patients will show improvement in regulation of physiological arousal in the autonomic nervous system relative to pretreatment.
3. To evaluate that hypothesis that symptoms associated with PTSD such as depression, anxiety, insomnia and quality of life will also be improved.
4. To evaluate the hypothesis that military veterans with PTSD can be successfully recruited into a yoga intervention study and will find the intervention acceptable and tolerable and will exhibit high compliance.

ELIGIBILITY:
Inclusion Criteria:

* Male and female military veterans and active duty military personnel aged 18 and older
* A DSM IV diagnosis of post-traumatic stress disorder
* Potential subjects on medications are eligible to participate in the study
* Potential subjects who receive ongoing medical or psychological treatment are eligible to participate in this study as long as these treatments do not include more than one hour weekly of relaxation and mind-body based stress reduction strategies (strategies directly related to meditation and yoga)
* Potential subjects are eligible to participate in this study if they have sufficient mental and physical ability to fully participate in the parameters of the study. Subjects must be able to understand and comply with instructions in the group yoga sessions and home practice, complete questionnaires, participate in clinical interviews, and take part in all data collection activities. Subjects with severe mental or physical concerns that may prevent them from understanding and/or complying with the treatment will be excluded. For example, potential subjects confined to wheelchairs will not be eligible, although subjects with artificial limbs who are able to reasonably participate in the intervention may be deemed eligible. These determinations will be made during discussions with potential subjects on a case by case basis during the screening process

Exclusion Criteria:

* Potential subjects are ineligible if pregnant and in their third trimester.
* Potential subjects are ineligible if they are confined to a wheel chair.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2009-08; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Clinician Administered PTSD Scale (CAPS) | pre-intervention and 10 weeks

SECONDARY OUTCOMES:
PTSD Checklist Military Version (PCL-M) | pre-intervention, 5 weeks, 10 weeks and 3 months post intervention
Impact of Events Scale - Revised (IES-R) | pre-intervention, 5 weeks, 10 weeks and 3 months post intervention
25-item Resilience Scale (RS) | pre-intervention, 5 weeks, 10 weeks and 3 months post intervention
Twenty-four-hour urinary samples | pre-intervention and 3 months post intervention
10-minute segment of a seated 30-minute electrocardiogram recording session | pre-intervention and 3 months post intervention
Beck Depression Inventory (BDI) | pre-intervention, 5 weeks, 10 weeks and 3 months post intervention
Spielberger State Trait Anxiety Inventory (STAI) | pre-intervention, 5 weeks, 10 weeks and 3 months post intervention
Daily Sleep Wake Diaries | during intervention (weeks 1-10) and 3 months post intervention
Quality of Life Enjoyment and Satisfaction Questionnaire (Q-LES-Q) | pre-intervention, 5 weeks, 10 weeks and 3 months post intervention
Credibility Expectancy Questionnaire (CEQ) | pre-intervention, 5 weeks, 10 weeks and 3 months post intervention
Body-Oriented State Questionnaire (BOSC) | pre-intervention, 5 weeks, 10 weeks and 3 months post intervention
5-Facet Mindfulness Questionnaire (FFMQ) | pre-intervention, 5 weeks, 10 weeks and 3 months post intervention
Perceived Stress Scale (PSS) | pre-intervention, 5 weeks, 10 weeks and 3 months post intervention
Yoga Follow-up Questionnaire | 3 months post intervention
PTSD Checklist Civilian Version (PCL-C) | pre-intervention, 5 weeks, 10 weeks and 3 months post intervention

CONTACTS AND LOCATIONS:
Overall Officials: Sat Bir S Khalsa, Ph.D., Principal Investigator — Brigham and Women's Hospital; Jennifer Johnston, MA, LMHC, Study Director — Northeastern University
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] van der Kolk BA, Roth S, Pelcovitz D, Sunday S, Spinazzola J. Disorders of extreme stress: The empirical foundation of a complex adaptation to trauma. J Trauma Stress. 2005 Oct;18(5):389-99. doi: 10.1002/jts.20047. PMID 16281237
- [Background] Hoge CW, Auchterlonie JL, Milliken CS. Mental health problems, use of mental health services, and attrition from military service after returning from deployment to Iraq or Afghanistan. JAMA. 2006 Mar 1;295(9):1023-32. doi: 10.1001/jama.295.9.1023. PMID 16507803
- [Background] Creamer M, Burgess P, McFarlane AC. Post-traumatic stress disorder: findings from the Australian National Survey of Mental Health and Well-being. Psychol Med. 2001 Oct;31(7):1237-47. doi: 10.1017/s0033291701004287. PMID 11681550
- [Background] van der Kolk BA. Clinical implications of neuroscience research in PTSD. Ann N Y Acad Sci. 2006 Jul;1071:277-93. doi: 10.1196/annals.1364.022. PMID 16891578
- [Background] Seligman MEP. Learned Optimism, 2nd Edition ed. New York, NY: Pocket Books; 1998.
- [Background] Morse DR, Cohen L, Furst ML, Martin JS. A physiological evaluation of the yoga concept of respiratory control of autonomic nervous system activity. Int J Psychosom. 1984;31(1):3-19. No abstract available. PMID 6590525